CLINICAL TRIAL: NCT00312663
Title: A Phase I/IIa Controlled Study of the Safety, Immunogenicity and Preliminary Efficacy of FMP011/AS01B Candidate Malaria Vaccine in Malaria-naive Adults Living in the United States
Brief Title: Phase I/II Trial of a Malaria Vaccine in Adults Living in the United States of America
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: GlaxoSmithKline (Industry); The PATH Malaria Vaccine Initiative (MVI) (Other); Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: WRAIR 1250; HSRRB A-13734 (Other: USAMRMC)
Record Dates: First submitted 2006-04-06; First posted 2006-04-10 (Estimated); Results first posted 2018-11-26 (Actual); Last update posted 2018-11-26 (Actual); Status verified 2018-05

CONDITIONS: Plasmodium Falciparum Malaria
Keywords: Vaccine; Phase I/II; Malaria; Liver Stage Antigen -1; Falciparum Malaria Protein -11; AS01B; adjuvant
MeSH Terms: conditions — Malaria, Falciparum; Malaria | interventions — AS01B adjuvant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 10ug dose FMP011 (Experimental): Falciparum Malaria Protein 11 with AS01B adjuvant
  Interventions: Biological: Falciparum Malaria Protein 11 with AS01B adjuvant.
- 50ug dose FMP011 (Experimental): Falciparum Malaria Protein 11 with AS01B adjuvant
  Interventions: Biological: Falciparum Malaria Protein 11 with AS01B adjuvant.

INTERVENTIONS:
Biological: Falciparum Malaria Protein 11 with AS01B adjuvant. — malaria experimental vaccine

SUMMARY:
Phase I/II Trial of a Malaria Vaccine, FMP011/AS01B, in Adults Living in the United States of America.

DETAILED DESCRIPTION:
* Controlled challenge, Phase I/IIa WRAIR study.
* Healthy, malaria-naive adults aged 18 - 50 years.
* 2 groups, 5 subjects in group A (10µg dose) and 13 subjects in group B(50µg dose).
* Control: none for immunization phase; infectivity controls for challenge and rechallenge phases. Six infectivity controls per day of challenge will be enrolled for the challenge phases, with 3 alternates available for challenge if needed.
* Vaccination schedule of 0, 1 months.
* Challenge of up to 13 subjects in Group B.
* Contingent upon short term efficacy, rechallenge of initially protected subjects 6 months (+/- 2 months) after second dose of vaccine.
* Self-contained study.
* Duration of the study, per subject: approximately 15 months (screening, enrollment, vaccination, challenge and rechallenge).
* Data collection will be by done onsite.

ELIGIBILITY:
Inclusion Criteria:

* A male or non-pregnant female 18 to 50 years of age (inclusive) at the time of screening.
* Written informed consent obtained from the subject before screening procedures.
* Free of obvious health problems as established by medical history and clinical examination before entering into the study.*
* Available to participate for duration of study (approximately 15 months).
* If the subject is female, she must be currently using birth control, must be surgically sterilized, or must be at least 1-year post menopausal.
* Pass a comprehension assessment test.

Exclusion Criteria:

* Prior receipt of an investigational malaria vaccine.
* Use of any investigational or non-registered drug or vaccine other than the study vaccine(s) within 28 days preceding the first dose of study vaccine, or planned use during the study period.
* Administration of chronic immunosuppressants or other immune modifying drugs within six months of vaccination.
* Chronic use of antibiotics with anti-malarial effects.
* Planned administration/ administration of a vaccine not foreseen by the study protocol within 30 days of the first dose of vaccine(s).
* History of use of anti-malarial medication within 60 days prior to vaccination.
* Any history of malaria.
* Known exposure to malaria within the previous 12 months.
* Planned travel to malarious areas during the study period.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including HIV infection.
* A family history of congenital or hereditary immunodeficiency.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Chronic or active neurologic disease including seizures, but not including a single febrile seizure as a child.
* History of splenectomy.
* Acute disease at the time of enrollment.
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory screening tests.
* Personal history of autoimmune disease or subjects who describe a first-degree relative with clearly documented autoimmune disease.
* Seropositive for hepatitis B surface antigen.
* Seropositive for Hepatitis C virus (antibodies to HCV).
* Administration of immunoglobulins and/or any blood products within the three months preceding the first dose of study vaccine or planned. administration during the study period
* Pregnant or lactating female.
* Suspected or known current alcohol abuse as defined by the American Psychiatric Association in DSM IV.
* Chronic or active intravenous drug use.
* History of severe reactions to mosquito bites as defined as anaphylaxis.
* Female who intends to become pregnant during the study.
* Any history of anaphylaxis in reaction to vaccination.
* A clinical history of sickle cell disease or sickle cell trait.
* Any other significant finding that in the opinion of the investigator would increase the risk of having an adverse outcome from participating in this study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2006-04; Primary Completion 2006-10 (Actual); Study Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James F. Cummings, MD, Principal Investigator — Walter Reed Army Institute of Research (WRAIR)
Locations (1):
- Walter Reed Army Institute of Research, Silver Spring, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
GlaxoSmithKline, The PATH Malaria Vaccine Initiative (MVI), Walter Reed Army Institute of Research (WRAIR)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 18 immunized subjects
Pre-assignment Details: 18 subjects were randomly assigned to the immunization phase for each of the 2 vaccine formulations.
Groups:
- Infectivity Controls (IC): 10 Subject from the high dose group and six non immunized subjects enrolled prior to challenge to serve as IC's for malaria sporozoite challenge.
Period: Immunization Phase
Arm/Group | 10ug Dose FMP011 | 50ug Dose FMP011 | Infectivity Controls (IC)
Started | 5 | 13 | 0
Completed | 5 | 12 | 0
Not Completed | 0 | 1 | 0
Not completed — Adverse Event | 0 | 1 | 0
Period: Challenge Phase
Arm/Group | 10ug Dose FMP011 | 50ug Dose FMP011 | Infectivity Controls (IC)
Started | 0 (low dose subjects didn't participate in the challenge phase) | 10 (10 subjects from the high dose group participated in the challenge phase) | 6 (6 non-immunized subjects participated in the challenge phase)
Completed | 0 | 10 | 6
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: 10 subjects from the high dose group and 6 non-immunized subjects participated in the Infectivity Control
Groups:
- Infectivity Control (IC): 10 Subject from the high dose group and six non immunized subjects enrolled prior to challenge to serve as IC's for malaria sporozoite challenge
- Total: Total of all reporting groups
Arm/Group | 10ug Dose FMP011 | 50ug Dose FMP011 | Infectivity Control (IC) | Total
Number analyzed (Participants) | 5 | 13 | 6 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.8 (7.9) | 32.8 (8.1) | 24.5 (4.9) | 32.2 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 8 | 0 | 9
  Male | 4 | 5 | 6 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 3 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 1 | 3
  White | 4 | 6 | 5 | 15
  More than one race | 0 | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 13 | 6 | 18

OUTCOME MEASURES:

1. Primary Outcome: Safety - Most Frequently Reported Adverse Events and Grade
Description: An AE was defined as any reaction, side effect, or untoward event that occurred during the course of the trial whether or not the event was considered related to the study drug or clinically significant. Grade 1: Mild Grade 2: Moderate Grade 3: Severe
Time Frame: 30 days post vaccination
Population: The AE's were tabulated and summarized by subject and treatment groups. No additional analyses were performed. Subjects from the IC group were not evaluated for AE's and there for not included in the data.
  Grade 1 = mild, Grade 2 = moderate, Grade 3 = severe
Measure: Number; unit: adverse events
Arm/Group | 10ug Dose FMP011 | 50ug Dose FMP011 | Infectivity Control (IC)
Number analyzed (Participants) | 5 | 13 | 0
adverse events
  Pain - Grade 1 | 5 | 9 |
  Pain - Grade 2 | 0 | 4 |
  Pain - Grade 3 | 0 | 0 |
  Redness - Grade 1 | 1 | 1 |
  Redness - Grade 2 | 1 | 1 |
  Redness - Grade 3 | 1 | 2 |
  Swelling - Grade 1 | 1 | 2 |
  Swelling - Grade 2 | 0 | 0 |
  Swelling - Grade 3 | 0 | 2 |

2. Secondary Outcome: Anti-LSA-1 Antibody Response in Titer Units on Days 0, 28, 42, and 84
Description: Anti-LSA-1 Antibody Response in Titer Units on Days 0, 28, 42, and 84
Time Frame: Days 0, 28, 42, and 84
Population: nAnti-LSA-1 Antibody Response in Titer units on Days 0, 28, 42 and 84
Measure: Median (Full Range); unit: Titer units
Arm/Group | 10ug Dose FMP011 | 50ug Dose FMP011 | Infectivity Controls (IC)
Number analyzed (Participants) | 5 | 13 | 6
Titer units
  Day 0 | 36.2 [23.7 to 644.0] | 43.15 [-10 to 475.9] | NA [NA to NA] — Didn't participate in phase
  Day 28 | 514.4 [51.9 to 3523.3] | 462.0 [41.1 to 6161.0] | NA [NA to NA] — Didn't participate in phase
  Day 42 | NA [NA to NA] — Didn't' participate in Challenge Phase | 36527.0 [1774.9 to 85080.0] | 21.1 [-10 to 248.5]
  Day 84 | NA [NA to NA] — Didn't' participate in Challenge Phase | 9180.0 [834.0 to 18131.0] | 30 [14.0 to 235.4]

ADVERSE EVENTS:
Time Frame: Up to 6 months
Description: Evaluate the safety by 1) occurrence of solicited AEs over a 7 day follow-up period (day of immunization and 6 days post-immunization); 2) the occurrence of unsolicited AEs over a 30 day follow-up period (day of immunization and 29 day follow-up period); and 3) the occurrence of SAEs during the study period. IC group was not included in AE evaluations and there for not reported in the FCSR.
Arm/Group | 10ug Dose FMP011 | 50ug Dose FMP011 | Infectivity Control (IC)
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/13 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/13 | 0/0
Other Adverse Events (participants affected / at risk) | 5/5 | 13/13 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 10ug Dose FMP011 (N=5) | 50ug Dose FMP011 (N=13) | Infectivity Control (IC) (N=0)
Pain (General disorders) | 5 (5) | 13 (13) | 0 (0) — Any
Swelling (General disorders) | 1 (1) | 4 (4) | 0 (0) — Any
Redness (Skin and subcutaneous tissue disorders) | 3 (3) | 4 (4) | 0 (0) — Any
Fever (General disorders) | 3 (3) | 5 (5) | 0 (0) — Any
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) — Any
Headache (Nervous system disorders) | 3 (3) | 10 (10) | 0 (0) — Any
Malaise (General disorders) | 3 (3) | 9 (9) | 0 (0) — Any
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 7 (7) | 0 (0) — Any
Fatigue (General disorders) | 2 (2) | 9 (9) | 0 (0) — Any
Joint pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4) | 0 (0) — Any
Pain (General disorders) | 5 (5) | 13 (13) | 0 (0) — Immunization 1
Swelling (General disorders) | 1 (1) | 2 (2) | 0 (0) — Immunization 1
Redness (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0) — Immunization 1
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) — Immunization 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) — Immunization 1
Fatigue (General disorders) | 1 (1) | 2 (2) | 0 (0) — Immunization 1
Joint pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) — Immunization 1
Pain (General disorders) | 4 (4) | 11 (11) | 0 (0) — Immunization 2
Swelling (General disorders) | 0 (0) | 3 (3) | 0 (0) — Immunization 2
Redness (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3) | 0 (0) — Immunization 2
Fever (General disorders) | 3 (3) | 5 (5) | 0 (0) — Immunization 2
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) — Immunization 2
Headache (Nervous system disorders) | 3 (3) | 9 (9) | 0 (0) — Immunization 2
Malaise (General disorders) | 3 (3) | 9 (9) | 0 (0) — Immunization 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 7 (7) | 0 (0) — Immunization 2
Fatigue (General disorders) | 2 (2) | 9 (9) | 0 (0) — Immunization 2
Joint pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4) | 0 (0) — Immunization 2
Chills (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 0 (0) — Any
Bruise (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) — Any
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) — Any
Flu-like symptoms (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) — Any
Stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) — Any
Swollen glands (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) — Any
Chills (Musculoskeletal and connective tissue disorders) | 2 (2) | 7 (7) | 0 (0) — Immunization 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) — Immunization 2
Flu-like symptoms (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) — Immunization 2
Stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) — Immunization 2
Swollen glands - neck and axillary (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) — Immunization 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No